CLINICAL TRIAL: NCT02105935
Title: Investigator Initiated Protocol for the: Evaluation of the Effectiveness and Clinical Utility of Brain Network Activation (BNA™) Technology in the Management of Sport Related Concussion and the Establishment of Normative Data in Youth and Adolescents Athletes.
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: ELM-23
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Normative; Concussed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normative study: male and female athletes, ages 8-14.
- Baseline: male and female athletes, ages 8-18.

SUMMARY:
This study's objectives are:

* To prospectively examine changes in brain network activation (BNA™) from baseline to recovery (i.e., return to activity) in youth and adolescent athletes with concussion.
* To assess the clinical utility of changes in BNA to assist in clinical decision-making.
* To generate normative BNA data.

DETAILED DESCRIPTION:
Currently, there is no direct, reliable, bed-side, and non-invasive method for assessing changes in brain activity associated with concussion. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a noninvasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA™) to temporally and spatially map brain function, connectivity and synchronization.

The proposed study will provide additional evidence for the utility and contribution of the BNA™ test (reflecting temporal and spatial changes in brain activity as well as brain functional connectivity associated with concussion) in concussion management.

ELIGIBILITY:
Inclusion Criteria:

* • Male and Female Athletes: Age 8-14 (Arm 1) or 8-18 years (Arm 2).

  * For Arm 1 - Over 3 days and below 7 days post-concussion (sports-related) and currently symptomatic
  * Able to speak, read and understand English sufficiently to understand the nature of the study, and to allow completion of all study assessments.
  * Willingness to participate and able to give informed assent (child) and Parental consent

Exclusion Criteria:

* Currently with lice or open wounds on scalp.
* Long and thick hair that prevents the proper administration of an EEG cap.
* Significant sensory deficits, e.g., deafness or blindness.

  * Normative Exclusion Criteria:
* Any chronic disease as determined by clinical evaluation and medical history.
* Any psychiatric disorder, e.g., depression, bipolar disorder, schizophrenic disorder, etc. as determined by clinical evaluation and the Mini International Neuropsychiatric Interview (MINI)
* Any CNS neurologic disorder, e.g., epilepsy, seizures, etc. as determined by clinical evaluation
* Any neuropsychological disorders, e.g.: ADHD, Autistic Spectrum Disorder (ASD), etc. as determined by clinical evaluation
* History of Special education, e.g., reading disorder (dyslexia), writing disorder (dysgraphia), math disorder (dyscalculia), nonverbal learning disorder.
* History of any medication affecting CNS within the last 3 months, e.g., antidepressants, anticonvulsants, psychostimulants, first generation antihistamines, etc.
* Substance abuse in the last 3 months.
* History of any clinically significant brain trauma as determined by the investigator.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: male and female athletes
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
quantitative and qualitative analysis of brain network activation (BNA) in participants that have sustained concussion compared to their baseline test. | 1 year
  quantitative and qualitative analysis of brain network activation (BNA) in participants that have sustained concussion compared to their baseline test.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Myer, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati children's hospital Sport center, Cincinnati, Ohio, United States